CLINICAL TRIAL: NCT00923819
Title: 4XL-Study - Obesity Surgery in Adolescence
Brief Title: 4XL Study - Obesity Surgery in Adolescence
Acronym: 4XL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset i Vestfold HF (Other)
Collaborators: The Hospital of Vestfold (Other)
Responsible Party: Principal Investigator, Samira Lekhal, PhD, MD, Sykehuset i Vestfold HF
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4XL-2009
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Obesity, Morbid
Keywords: Adolescents; Gastric Bypass; Quality of Life; Mental Health; Lifestyle
MeSH Terms: conditions — Obesity, Morbid; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Laparoscopic Gastric Bypass
  Interventions: Procedure: Laparoscopic gastric bypass
- Group B (Active Comparator): Standard conservative treatment. Patients from Child Obesity Registry of Vestfold.
  Interventions: Behavioral: Standard conservative treatment

INTERVENTIONS:
Procedure: Laparoscopic gastric bypass — Patients are referred to Morbid Obesity Center from Vestfold Hospital Trust and other hospitals in Norway. The procedure will take place at Morbid Obesity Center, Vestfold Hospital Trust.
  Arms: Group A
Behavioral: Standard conservative treatment — Participants from Child Obesity Registry who undergoes conservative treatment at Morbid Obesity Center, Vestfold Hospital Trust.
  Arms: Group B

SUMMARY:
The purpose of this study on adolescents between 13 and 18 years of age with morbid obesity is to determine whether surgical treatment gives more health benefits than standard conservative treatment, and if laparoscopic gastric bypass is a method with high safety and a low complication rate.

DETAILED DESCRIPTION:
The study has two intervention arms:

Experimental: Group A Surgery; laparoscopic gastric bypass

Active comparator: Group B Patients from Child Obesity Registry of Vestfold who get standard conservative treatment in a multidisiplinary team at Morbid Obesity Center.

All patients are referred to Morbid Obesity Center from other hospitals or general practionairs in Norway. The procedure will take place at the Vestfold Hospital Trust The participants are included for 2 years follow-up with visits to a multidisciplinary team every 3rd month at the Morbid Obesity Center. Total follow-up time is ten years.

ELIGIBILITY:
Inclusion Criteria:

* Between 13 and 18 years of age at inclusion
* Tanner stage 4-5
* BMI > 40 kg/m2 or BMI > 35 with at least one comorbidity (type 2-diabetes, obstructive sleep apnea, serious hypertension or cerebral pseudotumor)
* At least one year multidisciplinary treatment completed

Exclusion Criteria:

* Tanner stage < 4
* Substantial risk for lack of compliance
* Obesity syndrome (e.g., Prader Willi syndrome)
* Obesity related to brain damage
* Serious general disease
* Monogenic obesity

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-06 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
BMI and weight loss | Baseline, Year 1, 2, 5, 10
  Surgical or standard conservative treatment

SECONDARY OUTCOMES:
Quality of Life (KINDL) | 10 years
  Web-based questionnaire baseline and after 1, 2, 5 and 10 years.
Eating Disorders (Child Eating Behavior Questionnaire) | 10 years
  Web-based questionnaire baseline and after 1, 2, 5 and 10 years.
Mental Health (Development and Well-Being Assessment, DAWBA) | 10 years
  Web-based questionnaire baseline and after 1, 2, 5 and 10 years.
Self-Esteem (Rosenberg Self-Esteem scale) | 10 years
  Web-based questionnaire baseline and after 1, 2, 5 and 10 years.
Surgical and Medical Complications | 10 years
  Web-based questionnaire baseline and after 1, 2, 5 and 10 years.
Blood sample results | 10 years
  Blood tests are biobanked at baseline and after 1, 2, 5 and 10 years.

CONTACTS AND LOCATIONS:
Overall Officials: Samira Lekhal, PhD,MD, Principal Investigator — Vestfold Hospital Trust/The Hospital of Vestfold; Jøran Hjelmesæth, MD, PhD, Study Chair — Vestfold Hospital Trust/The Hospital of Vestfold
Locations (1):
- Morbid Obesity Center, The Hospital of Vestfold, South-Eastern Norway Regional Health Authority, Tønsberg, Norway